CLINICAL TRIAL: NCT00000990
Title: A Multicenter Placebo-Controlled Trial To Evaluate the Safety and Efficacy of Oral Zidovudine in the Treatment of Children Infected With Human Immunodeficiency Virus With Mild to Moderate Symptoms (Including LIP)
Brief Title: The Safety and Effectiveness of Zidovudine in the Treatment of HIV-Infected Children With Mild to Moderate Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 052; 11026 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pulmonary Fibrosis; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Pulmonary Fibrosis | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine the safety and usefulness of zidovudine (AZT) for the treatment of children 3 months to 12 years of age. This study is designed to determine if children who are infected with HIV and who have a special type of lung disease called lymphocytic interstitial pneumonitis (LIP) or other early symptoms of HIV infection may derive benefit from treatment with AZT. It is hoped that this drug will prevent children from developing additional symptoms and infections and will help resolve already existing symptoms.

AZT has been shown in the laboratory to inhibit the infection of cells by HIV. AZT has been shown to decrease the mortality and the frequency of opportunistic infections in certain adult patients with symptomatic HIV infection. It is, therefore, likely that symptomatic HIV-infected children may also benefit from specific antiviral therapy.

DETAILED DESCRIPTION:
AZT has been shown in the laboratory to inhibit the infection of cells by HIV. AZT has been shown to decrease the mortality and the frequency of opportunistic infections in certain adult patients with symptomatic HIV infection. It is, therefore, likely that symptomatic HIV-infected children may also benefit from specific antiviral therapy.

Children who participate in the study are evaluated at a hospital outpatient clinic and are under the care of a specialist in pediatrics. Of the children who participate in the study, half receive AZT syrup and half receive a placebo (sugar solution). The investigator does not know which medication each child receives as this is decided by a random process. The children take the medication in a strawberry-flavored clear syrup every 6 hours (4 times a day), for a period of 2 years or 104 weeks. The children are monitored on an outpatient basis while receiving therapy and the tests performed on admission to the study are repeated several times during treatment. Blood samples are obtained once a week for the first 4 weeks, every other week for the next 4 weeks, and then monthly until the end of the study. At certain sites, Cerebrospinal fluid (CSF) is collected by lumbar puncture every 52 weeks to evaluate infection involving the brain and nervous system. An independent committee reviews the data collected on the children every 6 months. The drug is stopped or the dose reduced if unacceptable side effects develop. AMENDED: As of August 7, 1989 the study blind was broken, the placebo arm discontinued and the study closed to accrual as of September 25, 1989. The 6 children enrolled in the study have been offered AZT.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis for Pneumocystis carinii pneumonia (PCP) in children with AIDS or CD4 cell count = or < 500 cells/mm3.

Children must demonstrate the following clinical and laboratory findings:

* Laboratory evidence of HIV infection as demonstrated by either a positive viral culture or detectable serum p24 antigen or = or > two positive tests for HIV antibody, which must be determined by a federally licensed ELISA test and confirmed by Western blot.
* Children < 15 months of age, who are thought to have acquired HIV through perinatal transmission and whose only laboratory evidence of HIV infection is a positive antibody test, must also have one or more of the following laboratory criteria indicative of immunologic abnormality:
* hypergammaglobulinemia (IgG or IgA) defined as greater than the upper limit of normal for age-adjusted normals; absolute depression in the CD4+ cells to = or < 500 cells/mm3; decreased helper/suppressor ratio < 1.0; depressed in vitro mitogen response to at least one antigen/mitogen.
* Absence of serious bacterial infections as defined in Exclusion Criteria requiring therapy at the time of entry.
* Hemophiliacs are included.

Exclusion Criteria

Co-existing Condition:

Children will be excluded for the following reasons:

* Recurrent or life-threatening toxicity. Several allergic reactions such as exfoliative erythroderma, anaphylaxis, or vascular collapse. The presence of one or more of the indicator diseases of AIDS, such as opportunistic infections, malignancy, recurrent bacterial infections, or encephalopathy. Development of two or more episodes of recurrent varicella zoster infection or chronic zoster defined as = or > 30 days duration. Development of AIDS related complex, with failure to thrive, persistent or recurrent oral candidiasis, plus at least one of the following:
* Diarrhea that is either persistent or recurrent, lymphadenopathy at two or more noncontiguous sites, organomegaly, nephropathy manifested by nephrotic syndrome without evidence of renal failure, two or more episodes of herpes stomatitis or one or more episodes of herpes zoster within a 1 year period; plus at least one of the following:
* hypergammaglobulinemia, depression in the CD4+ cells to = or < 500/mm3, decreased helper/suppressor ratio < 1.0, depressed in vitro mitogen response to at least one antigen/mitogen.

Concurrent Medication:

Excluded:

* Hepatotoxic drugs.
* Steroids for lymphocytic interstitial pneumonitis (LIP).
* Prophylaxis for oral candidiasis, or otitis media.
* Immunoglobulin therapy.
* Chronic use of drugs that are metabolized by hepatic glucuronidation.

Concurrent Treatment:

Excluded:

* Supplemental oxygen treatment for lymphocytic interstitial pneumonitis (LIP).

Children will be excluded from the study for the following reasons:

* AIDS-defining opportunistic infection or neoplasm.
* Unexplained recurrent, serious bacterial infections (= or > 2 within a 2-year period) including sepsis, meningitis, pneumonia, abscess of an internal organ, and bone/joint infections caused by Haemophilus, Streptococcus, or other pyogenic bacteria.
* Encephalopathy.
* One or both of the following:
* Failure to thrive, defined as a child who crosses two percentile lines on the growth chart or a child who is less than the fifth percentile and does not follow the curve; and/or persistent (= or > 2 months) oral candidiasis despite appropriate topical therapy.
* Children with lymphocytic interstitial pneumonitis (LIP) who are steroid dependent or requiring supplemental oxygen or who have a pretreatment PaO2 < 70 mmHg.
* Children who qualify for the entrance criteria to open-label zidovudine (AZT) or AZT plus or minus gammaglobulin.

Prior Medication:

Excluded:

* Rifampin or rifampin derivatives.
* Antiretroviral agents.
* Zidovudine (AZT).
* Excluded within 2 weeks of study entry:
* Other experimental therapy.
* Drugs which cause prolonged neutropenia or significant nephrotoxicity.
* Excluded within 4 weeks of study entry:
* Immunomodulating agents including immunoglobulin, interferon, isoprinosine, and IL-2.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Lymphocyte transfusions.

Active alcohol or drug abuse.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224
Dates: Study Completion 1992-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Weintrub, Study Chair
Locations (32):
- United States (32):
  - Kaiser Permanente / UCLA Med Ctr, Downey, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Martin Luther King Jr Gen Hosp / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Stanford Univ School of Medicine, Menlo Park, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSD Treatment Ctr, San Diego, California
  - Northern California Pediatric AIDS Treatment Ctr / UCSF, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Univ Babies' Hosp, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas